CLINICAL TRIAL: NCT00357890
Title: A Pilot Study of the Effect of Continuous Subcutaneous Insulin Infusion in Adolescents With Newly-diagnosed Type 1 Diabetes on Insulin Resistance, Beta-cell Function and the Honeymoon Period.
Brief Title: Insulin Pump Therapy in Adolescents With Newly Diagnosed Type 1 Diabetes (T1D)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Larry A. Fox, MD, Pediatric Endocrinologist, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-03890-002
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Insulin-Dependent
Keywords: type 1 diabetes; diabetes; new onset; CSII; insulin sensitivity; beta cell function; beta cell preservation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pump therapy (CSII) (Experimental): Use of pump therapy
  Interventions: Device: Insulin pump therapy
- Multiple daily injections (MDI) (Active Comparator): Use of MDI (basal bolus therapy with glargine)
  Interventions: Drug: Multiple daily injections using insulin glargine + rapid acting analog

INTERVENTIONS:
Device: Insulin pump therapy — CSII initiated within 1 month of diagnosis
  Other Names: Continuous subcutaneous insulin infusion (CSII)
  Arms: Pump therapy (CSII)
Drug: Multiple daily injections using insulin glargine + rapid acting analog — MDI as control
  Other Names: MDI using glargine plus a rapid acting analog
  Arms: Multiple daily injections (MDI)

SUMMARY:
Within 4 weeks after diagnosis of type 1 diabetes, 10 subjects (pubertal males, 12-17 years old) will be randomized to either receive multiple daily injection (MDI) using Lantus insulin, or continuous subcutaneous insulin infusion (CSII; pump therapy). The study evaluates how these modes of therapy affect insulin sensitivity (measured by the euglycemic-hyperinsulinemic clamp studies and adiponectin concentration changes) and beta cell function (measured by mixed meal tolerance testing).

DETAILED DESCRIPTION:
Within 4 weeks after diagnosis of type 1 diabetes, 10 subjects (pubertal males, 12-17 years old) will be randomized to either receive multiple daily injection (MDI) using Lantus insulin, or continuous subcutaneous insulin infusion (CSII; pump therapy). The proposed protocol compares the changes in diabetes control between pump therapy and MDI treatment groups. More importantly, however, the study evaluates how these modes of therapy may affect the honeymoon period and glycemic control, specifically focusing on changes in insulin sensitivity (measured by the euglycemic-hyperinsulinemic clamp studies and adiponectin concentration changes) and beta cell function (measured by mixed meal tolerance testing). Demonstrating that pump therapy at the time of diagnosis of type 1 diabetes prolongs the honeymoon phase by improving insulin sensitivity and beta cell function may have important therapeutic implications that could influence the standard of care in pediatric diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient between the age of 12 and 17 years inclusive at time of entry into study (i.e., after their 12th but before their 18th birthday)
* Type 1 diabetes mellitus for no more than 10 days
* pubertal (Tanner stage 2 or above)
* The patient and parents or guardians should be able to do simple math calculations (necessary for pump management)
* Parent or legal guardian must give signed informed consent

Exclusion Criteria:

* No other chronic medical conditions (well-controlled thyroid disease is OK, and mild asthma is OK if the patient is not on chronic inhaled or oral daily corticosteroids)
* Exceptional psychological stress, more than expected for circumstances of having the new diagnosis of diabetes
* Inability or unwillingness to comply with requirements of the protocol

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2005-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry A Fox, MD, Principal Investigator — Nemours Chidlren's Clinic
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pump Therapy (CSII) | Multiple Daily Injections (MDI)
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adolescents, 12-17 years old, with type 1 diabetes mellitus duration up to 10 days were enrolled. They were randomly assigned to either pump therapy (CSII group) or multiple daily injections (MDI group).
Groups:
- Total: Total of all reporting groups
Arm/Group | Pump Therapy (CSII) | Multiple Daily Injections (MDI) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (1.1) | 13.7 (1.4) | 13.9 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Insulin sensitivity - glucose infusion rate (GIR) obtained from hyperinsulinemic-euglycemic clamp. Higher GIR reflects higher insulin sensitivity, lower GIR reflects lower insulin sensitivity.
Time Frame: 24 months
Population: 12 adolescents were randomized, 6 per treatment group, well matched at baseline.
Measure: Mean (Standard Error); unit: mg/kg/min
Groups:
- Pump Therapy (CSII): Insulin pump therapy group
- Multiple Daily Injections (MDI): Control group - patients placed on multiple daily injections
Arm/Group | Pump Therapy (CSII) | Multiple Daily Injections (MDI)
Number analyzed (Participants) | 6 | 6
mg/kg/min
  Baseline | 8.6 (1.6) | 6.2 (1.3)
  24 month | 5.8 (1.0) | 4.8 (0.9)

2. Primary Outcome: Beta Cell Function
Description: Beta cell function as assessed by peak c-peptide using mixed meal tolerance testing
Time Frame: 24 months
Population: 12 adolescents were randomized, 6 per treatment group, well matched at baseline.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Pump Therapy (CSII) | Multiple Daily Injections (MDI)
Number analyzed (Participants) | 6 | 6
ng/mL
  Baseline | 2.1 (0.4) | 1.7 (0.3)
  24 months | 1.1 (0.4) | 1.6 (0.9)

3. Secondary Outcome: Hemoglobin A1c
Description: Hemoglobin A1c (HbA1c) (%)
Time Frame: 24 months
Population: 12 adolescents were randomized, 6 per treatment group, well matched at baseline.
Measure: Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Groups:
- Multiple Daily Injections (MDI): Multiple daily injections group - patients placed on standard therapy with MDI
Arm/Group | Pump Therapy (CSII) | Multiple Daily Injections (MDI)
Number analyzed (Participants) | 6 | 6
percentage of glycosylated hemoglobin
  Baseline | 10 (0.4) | 10.2 (0.3)
  12 months | 6.1 (0.3) | 7.0 (0.6)
  24 months | 6.8 (0.4) | 7.5 (0.5)

4. Secondary Outcome: Percent Body Fat
Description: Percent body fat based on DEXA scan (%BF)
Time Frame: 24 months
Population: 12 adolescents were randomized, 6 per treatment group, well matched at baseline.
Measure: Mean (Standard Error); unit: percentage of body fat
Groups:
- Pump Therapy (CSII): Insulin pump therapy group - participants placed on CSII
Arm/Group | Pump Therapy (CSII) | Multiple Daily Injections (MDI)
Number analyzed (Participants) | 6 | 6
percentage of body fat
  Baseline | 20 (2.6) | 21.6 (4.0)
  12 months | 18.5 (3.6) | 20.3 (3.8)
  24 months | 17.4 (2.5) | 20.5 (2.3)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Pump Therapy (CSII) | Multiple Daily Injections (MDI)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
Pilot study and thus sample size is small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes